CLINICAL TRIAL: NCT02787486
Title: A Clinical Study to Evaluate the Relative Clinical Sensitivity, Specificity, and Performance of the a Laboratory Developed Test as a Screening Test for Fetal Chromosomal Aneuploidy, Infectious and Other Diseases, and RhD Genotyping in the General Population of Pregnant Women
Brief Title: Expanded Noninvasive Genomic Medical Assessment: The Enigma Study
Status: Completed | Type: Observational
Sponsor: Progenity, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-102-ENIGMA
Record Dates: First submitted 2016-05-26; First posted 2016-06-01 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-01

CONDITIONS: Down Syndrome; Edwards Syndrome; Patau Syndrome; Klinefelter Syndrome; Turner Syndrome; DiGeorge Syndrome; Chromosome Deletion; Aneuploidy
Keywords: Down syndrome; Edwards syndrome; Patau syndrome; Klinefelter syndrome; DiGeorge syndrome; Chromosome Deletion; Aneuploidy
MeSH Terms: conditions — Down Syndrome; Trisomy 18 Syndrome; Trisomy 13 Syndrome; Klinefelter Syndrome; Turner Syndrome; DiGeorge Syndrome; Chromosome Deletion; Aneuploidy | interventions — Blood Specimen Collection; Telbivudine

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Aneuploidy Arm: Includes pregnant women at high risk for fetal chromosome aneuploidy for serum screening
  Interventions: Other: Blood sampling for Laboratory Developed Test (LDT) analysis
- TORCH Arm: Infectious disease arm: Toxoplasmosis, other viruses, rubella, cytomegalovirus, and herpes simplex virus (TORCH). Includes pregnant women at low-risk for fetal aneuploidy that may be at increased risk for fetal infection for serum screening
  Interventions: Other: Blood sampling for Laboratory Developed Test (LDT) analysis

INTERVENTIONS:
Other: Blood sampling for Laboratory Developed Test (LDT) analysis — Each enrolled subject, either in the first or second trimester, will donate up to 50 mL (just over 3 tablespoons) of whole blood for development of the LDT

SUMMARY:
In January 2007, the American Congress of Obstetricians and Gynecologists (ACOG) revised its guidelines that now recommend physicians are ethically obligated to fully inform all pregnant women that screening for fetal chromosomal abnormalities including biochemical screening tests and invasive procedures such as CVS or amniocentesis is available, regardless of age. Further, it is entirely up to the patient to decide whether or not she wishes to be screened for fetal chromosomal abnormalities without judgment from the physician.

Noninvasive laboratory-developed tests (LDTs) that detect an abnormal amount of maternal and fetal DNA in an expectant mother's blood sample (known as circulating cell-free DNA) are now available. These LDTs have not been cleared or approved by the U.S. Food and Drug Administration (FDA). Although LDTs to date have not been subject to U.S. FDA regulation, certification of the laboratory is required under the Clinical Laboratory Improvement Amendments (CLIA) to ensure the quality and validity of the test.

To sample collection study will obtain whole blood specimens from pregnant subjects to be used for development of prenatal assays to assist in the screening for fetal genetic abnormalities, infectious and other diseases, and blood group typing through detection of circulating cell-free DNA extracted from maternal plasma.

DETAILED DESCRIPTION:
Eligible subjects will provide written informed consent after which basic demographic and clinical data will be collected.

Study procedures involve the collection of 50 mL of whole blood at one or more monthly clinic visits (≥25 days apart) from pregnant women (18 to 54 yrs of age) carrying a single fetus of 8 to 22 weeks of gestational age inclusive.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing to provide informed consent and comply with study procedures
* Pregnant female, 18 to 54 years of age carrying a singleton fetus of 8 to 22 weeks gestational age
* Willing to provide a study blood sample in accordance with the protocol
* Willing to allow access to her medical records to collect pregnancy outcome information
* Willing to provide consent for release of fetal karyotype if an invasive procedure (CVS or amniocentesis) is performed during the pregnancy
* Subject is known to be at risk for one or more of the following:
* fetal gene and chromosome abnormalities (e.g., T21, T18, T13, microdeletion syndromes, sex chromosome abnormalities)
* congenital fetal infection (e.g. toxoplasmosis, syphilis, HIV, rubella, CMV, HSV)
* irregular blood group antigens (subject or father of the baby)
* other condition amenable to noninvasive prenatal testing such as a single gene disorder (e.g., CF, sickle cell, Fragile X)

Exclusion Criteria:

* No fetal heart activity detected
* Mother or father have known chromosomal abnormalities (including known balanced translocations)
* Women with active or history of malignancy

Ages: 18 Years to 54 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All pregnant women undergoing standard maternal serum screening for fetal aneuploidy will be considered for enrollment as well as those with a priori risk factors for fetal aneuploidy.
Sampling Method: Non-Probability Sample
Enrollment: 760 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Point estimates and 95% CIs for sensitivity, specificity, PPV, and NPV versus birth outcome (trisomy or Unaffected/non-trisomy) for the LDT in the population of pregnancies at mixed-risk for chromosomal abnormalities | about 3 years
  Primary Objective

SECONDARY OUTCOMES:
To estimate the false positive rate of the LDT versus birth outcome (trisomy or Unaffected/ non-trisomy) in a low-risk sub-population of pregnant women undergoing serum biochemical screening for fetal aneuploidy. | about 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Stiegler, PhD, Study Director — Head of Clinical Affairs
Locations (8):
- United States (8):
  - Valley Perinatal, Scottsdale, Arizona
  - Heinen Obstectrics & Gynecology, Eunice, Louisiana
  - Newlife Wellness OBGYN, Brooklyn, New York
  - Lakeshore Women's Specialists, Mooresville, North Carolina
  - Cincinnati Obgyn, Cincinnati, Ohio
  - James D. Kasten, M.D., Inc., Norwalk, Ohio
  - Regional Obstetrical Consultants, Chattanooga, Tennessee
  - Texas Maternal-Fetal Medicine, Webster, Texas

IPD SHARING:
Plan to Share IPD: Undecided